CLINICAL TRIAL: NCT00122044
Title: Childhood Hypertonia of Central Origin: An Open Label Trial of Anticholinergic Treatment Effects
Brief Title: Childhood Hypertonia of Central Origin: A Trial of Anticholinergic Treatment Effects
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Southern California (Other)
Collaborators: United Cerebral Palsy Foundation (Other); Don and Linda Carter Foundation (Other); Crowley Carter Foundation (Other)
Responsible Party: Principal Investigator, Terence Sanger, Associate Professor, University of Southern California
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CHOCOLATE
Record Dates: First submitted 2005-07-18; First posted 2005-07-21 (Estimated); Last update posted 2014-05-23 (Estimated); Status verified 2014-05

CONDITIONS: Dystonia
Keywords: childhood; cerebral palsy; dystonia; secondary; trihexyphenidyl; pediatric dystonia
MeSH Terms: conditions — Dystonia; Cerebral Palsy; Neoplasm Metastasis | interventions — Trihexyphenidyl

INTERVENTIONS:
Drug: trihexyphenidyl

SUMMARY:
This study is an open-label trial of trihexyphenidyl in children with upper extremity dystonia due to cerebral palsy. It is hypothesized that trihexyphenidyl in doses up to 0.75mg/kg/day would be well-tolerated and show significant changes on the Melbourne scale of upper extremity function.

DETAILED DESCRIPTION:
BACKGROUND: Although trihexyphenidyl has been used to treat both primary and secondary dystonia in children, previous studies have not investigated efficacy in secondary dystonia. We describe the results of a prospective, open-label, multi-center trial of high-dose trihexyphenidyl in children with secondary dystonia of the arms due to cerebral palsy.

METHODS: Twenty-six children age 4-15 years with cerebral palsy and dystonia that impairs function of the dominant upper extremity were enrolled. All children were given trihexyphenidyl at increasing doses over 9 weeks up to 0.75mg/kg/day. Trihexyphenidyl was subsequently tapered over 5 weeks. Visits occurred at baseline, 9 weeks, and 15 weeks. The primary outcome measure was the Melbourne assessment of upper extremity function, tested in the dominant arm.

RESULTS: Three children withdrew due to non-serious adverse events (chorea, drug rash, hyperactivity). 3 children reduced dosage due to non-serious adverse events. The 23 children who completed the study showed a significant improvement in arm function at 15 weeks (p=0.045) but not at 9 weeks. Post-hoc analysis showed that a subgroup (N=10) with hyperkinetic dystonia worsened at 9 weeks (p=0.04) but subsequently returned to baseline following taper of the medicine.

CONCLUSIONS: Trihexyphenidyl appears to be safe and effective for treatment of arm dystonia in children with cerebral palsy. Children with hyperkinetic dystonia may worsen. A larger randomized prospective trial is needed to confirm these results.

ELIGIBILITY:
Inclusion Criteria:

* Dystonia in the dominant upper extremity

Exclusion Criteria:

* Complete absence of voluntary movement in the affected hands, wrists, and elbows
* Severe weakness in the dominant upper extremity (MRC grade < 4)
* Passive range of motion at the hand, wrist or elbow less than 80% of normal
* Current use of medications for dystonia (anticholinergics, L-dopa, baclofen, diazepam, tizanidine, tetrabenazine, reserpine, and others)
* Changes in the subject's physical therapy regimen for the duration of the 15-week study
* Prior use of trihexyphenidyl or other anticholinergic therapy for dystonia.
* History of surgery on the dominant upper extremity or cervical spine
* Botulinum toxin injection in the dominant upper extremity within the previous 6 months
* Current or prior implantation of an intrathecal baclofen pump, deep brain stimulator, or other device to treat dystonia or spasticity
* Concurrent acute or chronic medical condition (such as frequent seizures, heart disease, or asthma) that could adversely affect motor performance or the safety of testing
* Presence of diurnal fluctuations or other clinical signs and symptoms suggesting an inborn error of metabolism, a family history of dystonia suggesting a genetic dystonia, or dystonia due to injury after the neonatal period (including toxin exposure, trauma, or medication-induced)
* History of allergic or adverse reaction to trihexyphenidyl or other anticholinergic medications
* Current complaint of urinary retention requiring treatment.
* History of glaucoma, or family history of glaucoma with onset before age 40

Ages: 5 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 35
Dates: Start 2003-01; Primary Completion 2004-12 (Actual); Study Completion 2004-12

PRIMARY OUTCOMES:
Melbourne assessment of upper extremity function

SECONDARY OUTCOMES:
Barry-Albright Dystonia Scale
Burke-Fahn-Marsden Dystonia Scale
Pediatric Outcomes Data Collection Instrument
Pediatric Quality of Life
Gross Motor Function Measure

CONTACTS AND LOCATIONS:
Overall Officials: Terence D Sanger, MD, PhD, Principal Investigator — Stanford University
Locations (7):
- United States (7):
  - University of Alabama School of Medicine, Birmingham, Alabama
  - Stanford University, Stanford, California
  - Rehabilitation Institute of Chicago, Chicago, Illinois
  - Kennedy Krieger Institute, Baltimore, Maryland
  - Washington University School of Medicine, St Louis, Missouri
  - University of Rochester Medical Center, Rochester, New York
  - Texas Scottish Rite Hospital for Children, Dallas, Texas

REFERENCES:
- See also: Information on childhood dystonia and other movement disorders — http://www.kidsmove.org